CLINICAL TRIAL: NCT07195812
Title: Evaluation of the Efficacy and Safety of Rivaroxaban in Improving Slow Coronary Flow After Percutaneous Coronary Intervention in STEMI Patients: A Multicenter, Prospective,Randomized, Controlled Study
Brief Title: Rivaroxaban for Slow Coronary Flow After PCI in STEMI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Affiliated Hospital of Jiaxing University (Other); The Second Affiliated Hospital of Jiaxing University (Other); Wenzhou People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20251206
Record Dates: First submitted 2025-09-17; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: ST Elevation Myocardial Infarction; No-Reflow Phenomenon
Keywords: Rivaroxaban; ST Elevation Myocardial Infarction; Slow Coronary Flow; No-Reflow Phenomenon; Antiplatelet Therapy; Percutaneous Coronary Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction; No-Reflow Phenomenon | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Therapeutics; Rivaroxaban; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Antiplatelet Therapy (Active Comparator): DAPT (aspirin 100 mg daily plus clopidogrel 75 mg daily or ticagrelor 90 mg per dose, twice daily) for 30 consecutive days
  Interventions: Drug: Dual Antiplatelet (DAPT) Therapy
- Rivaroxaban (Experimental): Rivaroxaban (2.5 mg twice daily) plus aspirin 100 mg daily plus clopidogrel 75 mg daily for 30 days
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Dual Antiplatelet (DAPT) Therapy — aspirin 100 mg daily plus clopidogrel 75 mg daily or ticagrelor 90 mg per dose, twice daily for 30 consecutive days
  Other Names: DAPT
  Arms: Dual Antiplatelet Therapy
Drug: Rivaroxaban — Rivaroxaban (2.5 mg twice daily) plus aspirin 100 mg daily plus clopidogrel 75 mg daily for 30 days
  Other Names: Rivaroxaban + Aspirin + Clopidogrel
  Arms: Rivaroxaban

SUMMARY:
The goal of this clinical trial is to learn if drug Rivaroxaban works to improve slow flow in STEMI patients after PCI in adults. It will also learn about the safety of drug Rivaroxaban. The main questions it aims to answer are:

Does drug Rivaroxaban Reduce the Corrected TIMI Frame Count (cTFC) in 1 Week After PCI ?

Researchers will compare Combination therapy with rivaroxaban (2.5 mg administered twice daily), aspirin (100 mg administered daily), and clopidogrel (75 mg administered daily) to Dual Antiplatelet Therapy to see if drug Combination therapy with rivaroxaban, aspirin works to treat Slow Flow in STEMI Patients After PCI.

Participants will:

Take drug Combination therapy with rivaroxaban (2.5 mg administered twice daily), aspirin (100 mg administered daily), and clopidogrel (75 mg administered daily) or Dual Antiplatelet Therapy every day for 1 months.

Visit the clinic in 7 days、30 days and 365 days for checkups and tests.

DETAILED DESCRIPTION:
The trial is a multicenter, prospective, randomized, open-label, controlled, pilot trial evaluating the efficacy and safety of rivaroxaban for improving slow coronary flow in ST-segment elevation myocardial infarction (STEMI) patients after percutaneous coronary intervention (PCI). Patients with STEMI who have undergone PCI and exhibit slow coronary flow (TIMI flow grade >0，and < 3, ) are eligible for the clinical trial. Slow coronary flow will be quantitatively assessed using the corrected TIMI frame count (cTFC) method.

The study consists of two parallel treatment groups, evaluating the clinical efficacy and safety of 30 days of combination antithrombotic therapy versus standard therapy, followed up to 365 days. The treatment groups are:

Group 1 - Experimental Antithrombotic Therapy Eligible patients will receive a combination of rivaroxaban (2.5 mg orally twice daily) plus dual antiplatelet therapy (DAPT: aspirin 100 mg/day and clopidogrel 75 mg/day) for a total duration of 30 days (treatment period), followed by assessments at 7 days, 30 days, and 365 days (follow-up period).

Group 2 - Standard Antithrombotic Therapy (Control) Eligible patients will receive standard DAPT (aspirin 100 mg/day and clopidogrel 75 mg/day or ticagrelor 90 mg twice daily) for a total duration of 30 days (treatment period), followed by assessments at 7 days, 30 days, and 365 days (follow-up period).

The primary efficacy endpoint is the change in cTFC from baseline to within 1 week after PCI. Key secondary endpoints include the incidence of Major Adverse Cardiovascular Events (MACE) and bleeding events (assessed by BARC criteria) at 7 days, 30 days, and 365 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, regardless of gender;
* Patients with ST-segment elevation myocardial infarction (STEMI) (meeting the diagnostic criteria of the 2019 Chinese "Guidelines for the Diagnosis and Treatment of Acute ST-Segment Elevation Myocardial Infarction");
* Patients undergoing percutaneous coronary intervention (PCI);
* Patients with slow flow after PCI (TIMI flow grade > 0 but < 3);
* Signed informed consent form and willingness to comply with follow-up.

Exclusion Criteria:

* Presence of malignant tumors or diseases with a life expectancy of less than 1 year;
* Coagulation disorders, diagnosed or suspected hematological diseases (excluding mild or moderate anemia);
* Thrombocytopenia (platelet count < 100 × 10⁹/L); history of severe gastrointestinal diseases or peptic ulcers; active bleeding within the past 3 months or major surgery history; history of intracranial hemorrhage or intracranial aneurysm;
* History of cerebral hemorrhage or ischemic stroke within the past 6 months;
* Patients with cardiogenic shock; systemic infections or immune system diseases; confirmed, highly suspected, or unable to rule out aortic dissection; severe uncontrolled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 110 mmHg);
* Current use of rivaroxaban or requiring long-term anticoagulation therapy (e.g., atrial fibrillation);
* Patients with renal insufficiency (eGFR < 15 mL/min/1.73m²) or hepatic insufficiency (Child-Pugh Class B or C);
* Lactating or pregnant women, or women of childbearing potential unable to use effective contraception during the study period;
* Patients with any contraindications or allergies to rivaroxaban, aspirin, clopidogrel, or ticagrelor;
* Participation in other clinical trials within the past 3 months;
* Other conditions deemed unsuitable for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change in Corrected TIMI Frame Count (cTFC) from baseline within 1 week after PCI | Change from baseline within 1 week
  Angiographic image acquisition should be standardized to a frame rate of 30 frames per second (fps). The TIMI frame count is calculated by determining the number of frames required for the contrast agent to travel from the initial opacification of the vessel to a standardized distal landmark. The designated distal landmarks vary depending on the coronary artery branch: for the left anterior descending artery (LAD), it is the distal bifurcation; for the left circumflex artery (LCx), it is the most distal branch of the obtuse marginal artery; and for the right coronary artery (RCA), it is the first branch of the posterolateral artery. Due to the longer length of the LAD compared to the LCx and RCA, the frame count for the LAD is divided by 1.7 to correct for this difference. The resulting value is the cTFC.

SECONDARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) and bleeding events | Assessed at 7 days, 30 days, and 365 days post-Percutaneous Coronary Intervention (PCI).
  The incidence of Major Adverse Cardiovascular Events (MACE), defined as a composite of Non-fatal myocardial infarction, cardiac death, stroke, target vessel revascularization, and stent thrombosis, and the incidence of bleeding events, classified according to the Bleeding Academic Research Consortium (BARC) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Jiang, Doctor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University

IPD SHARING:
Plan to Share IPD: No